CLINICAL TRIAL: NCT02242032
Title: A Double-Masked, Randomized, Placebo-Controlled Dose Escalation Study of the Safety and Tolerability of P 321 Ophthalmic Solution in Subjects With Dry Eye Disease
Brief Title: Study of the Safety and Tolerability of P 321 Ophthalmic Solution in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parion Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-321-101
Record Dates: First submitted 2014-08-28; First posted 2014-09-16 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-05

CONDITIONS: Dry Eye Disease
Keywords: dry eye disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- P-321 (Experimental): P-321 Ophthalmic Solution
  Interventions: Drug: P-321 Ophthalmic Solution
- P-321 Ophthalmic Solution Placebo (Placebo Comparator): P-321 Ophthalmic Solution Placebo
  Interventions: Drug: P-321 Ophthalmic Solution placebo

INTERVENTIONS:
Drug: P-321 Ophthalmic Solution
  Other Names: P-321
  Arms: P-321
Drug: P-321 Ophthalmic Solution placebo — Placebo to match P-321 Ophthalmic Solution
  Other Names: placebo
  Arms: P-321 Ophthalmic Solution Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of P-321 Ophthalmic Solution in subjects with mild to moderate dry eye disease.

DETAILED DESCRIPTION:
This is a single-center, dose escalation, randomized, double-masked, placebo-controlled, Phase 1/2a trial designed to evaluate the safety and tolerability of P-321 Ophthalmic Solution in subjects with mild to moderate dry eye for up to 4-weeks of treatment and up to 8 scheduled in clinic visits. This study will conduct a consecutive dose escalation of the following concentrations of P-321 Ophthalmic Solution given two times a day via ocular instillation: 0.0005% (Cohort 1), 0.0015% (Cohort 2), 0.005% (Cohort 3), and 0.01% (Cohort 4). Up to 48 subjects will be enrolled in four consecutive cohorts. Subjects will be randomized to P-321 Ophthalmic Solution or placebo in a 3:1 ratio.

Safety and tolerability assessments, drug plasma concentrations and drug urine concentrations will be evaluated throughout the study in all cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both genders and any race will be eligible for study participation if they:

  1. Provide written informed consent.
  2. Are 18 - 80 years of age.
  3. Corneal fluorescein staining score ≥2/15 on the NEI/Industry scale
  4. Conjunctival lissamine staining score of ≥ 2/18 on the NEI/Industry scale
  5. Schirmer <10mm/5min
  6. Are willing and able to follow instructions and can be present for the required study visits for the duration of the study.
  7. Female patients of child bearing potential must have a negative urine pregnancy test at Screening and agree to use a medically acceptable form of birth control. Male subjects who are sexually active must be willing to use highly effective contraception (i.e., less than 1% failure rate) during heterosexual intercourse from Day 1 through completion of the study.
  8. Have a history of Dry Eye Disease in both eyes supported by a previous clinical diagnosis or have a self-reported history of subjective complaints for at least 4 months prior to Screening, low tear volume, and ocular staining.
  9. Have documented history of topical lubricants at least daily or the desire to use topical lubricants in the past 4 months.
  10. Have normal lid anatomy

Exclusion Criteria:

* Individuals are not eligible for study participation if:

  1. Have anterior segment eye disease except primary dry eye.
  2. Patients with an identifiable or suspected secondary dry eye, i.e., a documented or likely systemic, ocular, pharmacologic, post-traumatic, post-surgical, or external cause for dry eye symptoms or ocular surface staining.
  3. Patients with current punctal plugs, punctal occlusion, or history of nasolacrimal duct obstruction are excluded.
  4. Have a history of glaucoma or intraocular pressure (IOP) > 25 mmHg at the Screening Visit (Visit 1) or a history of elevated IOP within the past year prior to Visit 1
  5. Contact lenses wear in the previous 30 days or during the Treatment Phase of the study.
  6. Use of lid scrubs (including baby shampoos)
  7. Known hypersensitivity to the study investigational medicinal product, or formulation excipients, including amiloride or related drugs or allergies to the components of the study drug.
  8. Any significant chronic illness that, in the opinion of the Principal Investigator (PI), could interfere with the study parameters.
  9. Use of any investigational product or device within 30 days prior to the Screening Visit or during the study.
  10. Those unable in the opinion of the PI to comply fully with the study requirements or complete the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Days 0, 1, 2, 8, 15, 22 and 28
  One primary objective of this trial is to assess the safety of P-321 Ophthalmic Solution versus placebo in subjects with moderate dry eye disease at 14 days (Cohorts 1-4) and 28 days (Cohort 4 only).
Changes from baseline in 14 days in visual acuity. | Change from baseline at 14 days.
  Change from baseline at 14 days in visual acuity.
Change from baseline at 28 days in visual acuity for Cohort 4 only. | Change from baseline at 28 days in visual acuity.
  Change from baseline at 28 days in visual acuity for Cohort 4 only.
Changes from baseline at 14 days in corneal staining. | Changes from baseline at 14 days.
  Changes from baseline at 14 days in corneal staining.
Changes from baseline at 28 days in corneal staining for cohort 4 only. | Changes from baseline at 28 days.
  Changes from baseline at 28 days in corneal staining for cohort 4 only.
Changes from baseline at 14 days in conjunctival staining. | Changes from baseline at 14 days
  Changes from baseline at 14 days in conjunctival staining.
Changes from baseline at 28 days in conjunctival staining for Cohort 4 only. | Changes from baseline at 28 days
  Changes from baseline at 28 days in conjunctival staining for Cohort 4 only.
Changes from baseline at 14 days in intraocular pressure. | Changes from baseline at 14 days.
  Changes from baseline at 14 days in intraocular pressure.
Changes from baseline at 28 days in intraocular pressure. for Cohort 4 only. | Changes from baseline at 28 days
  Changes from baseline at 28 days in intraocular pressure. for Cohort 4 only.
Changes from baseline at 14 days in ophthalmoscopy. | Changes from baseline at 14 days
  Changes from baseline at 14 days in ophthalmoscopy.
Changes from baseline at 28 days in ophthalmoscopy for Cohort 4 only. | Changes from baseline at 28 days
  Changes from baseline at 28 days in ophthalmoscopy for Cohort 4 only.

SECONDARY OUTCOMES:
Measure plasma P-321 concentrations | Pre-dose 0.5, 1, 2, 4, and 6 hours post dosing on Days 1 and Day 15 and pre-dose on Day 8.
  Drug plasma concentrations will be evaluated pre-dose 0.5, 1, 2, 4, and 6 hours post dosing on Days 1 and 15 and pre-dose on Day 8.
Measure urine concentrations of P-321 | At multiple timepoints throughout the study
  Drug urine concentrations will be evaluated at Day 1 and Day 15.
Measure tear concentrations of P-321 | pre-dose 0.5, 1, 2, 4, and 6 hours post dosing on Day 1 and Day 15 and pre-dose on Day 8.
  Drug tear concentrations will be evaluated at all visits post dose.
Measure plasma P-321 concentrations in Cohort 4 | pre-dose on Day 8 and Day 22, and pre-dose, 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose on Day 28
  Measure plasma P-321 concentrations in Cohort 4
Measure urine concentrations of P-321 in Cohort 4 | Day 28
  Measure urine concentrations of P-321 in Cohort 4
Measure tear concentrations of P-321 in Cohort 4 | pre-dose on Day 8 and Day 22, and pre-dose, 0.5, 1, 2, 4, 6, 8, and 24 hours post-dose on Day 28
  Measure tear concentrations of P-321 in Cohort 4

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Sall, MD, Principal Investigator — Sall Research Medical Center
Locations (1):
- Sall Research Medical Center, Artesia, California, United States